CLINICAL TRIAL: NCT05154058
Title: Dissection Technique of Medial Subperiosteal Release on the Incidence of Pes Bursitis
Brief Title: Medial Peel Release Technique TKA Randomized Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study was terminated due to principal investigator moving institutions
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ajay Premkumar, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003277
Record Dates: First submitted 2021-11-23; First posted 2021-12-10 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis, Knee
Keywords: Medial Subperiosteal Release
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: electrocautery (Active Comparator): Primary patients with Osteoarthritis (OA) undergoing Total Knee arthroplasty (TKA) will be randomly assigned into either the control or investigational group. The control arm of the study will undergo medial sub periosteal release with electrocautery.
  Interventions: Procedure: Medial Subperiosteal Release with Electrocautery
- Investigational: sharp dissection. (Active Comparator): Primary patients with OA undergoing TKA will be randomly assigned into either the control or investigational group. The investigational arm will undergo medial sub periosteal release using sharp dissection.
  Interventions: Procedure: Medial Subperiosteal Release with Sharp Dissection

INTERVENTIONS:
Procedure: Medial Subperiosteal Release with Sharp Dissection — Medial subperiosteal release - a routine step during primary total knee arthroplasty that will be conducted on every enrolled patient. This is commonly performed both via scalpel (aka sharp medial peel) or electrocautery
  Other Names: Medial Peel
  Arms: Investigational: sharp dissection.
Procedure: Medial Subperiosteal Release with Electrocautery — Medial subperiosteal release - a routine step during primary total knee arthroplasty that will be conducted on every enrolled patient. This group will receive this procedure using electrocautery.
  Arms: Control: electrocautery

SUMMARY:
Medial subperiosteal release is a commonly performed technique to improve surgical exposure and aid in joint balancing. This is a routine step during primary total knee arthroplasty that will be conducted on every enrolled patient. This is commonly performed both via scalpel (aka sharp medial peel) or electrocautery. The intervention will be randomly assigning subjects undergoing TKA into two groups, one receiving subperiosteal release using a scalpel (aka sharp medial peel) and the other via electrocautery.

DETAILED DESCRIPTION:
Medial release is a commonly performed technique to improve surgical exposure and aid in joint balancing. It is thought to be linked to the postoperative incidence of pes bursitis. However, the effect of scalpel vs electrocautery techniques for subperiosteal release has not been examined for their potential effect on the rates of pes bursitis. This randomized clinical trial will assign patients undergoing TKA for osteoarthritis (OA) into either scalpel or electrocautery release groups for their operation and will be followed postoperatively at 3 weeks and 3,6, and 12 months in order to determine the effect of release technique on rates of pes bursitis. This study will take place at Emory Orthopaedics. Subjects will not be compensated. Patients presenting to the clinic for evaluation of TKA will be screened for their eligibility in this study and recruited as well as consented in the clinic. This study can advance current clinical knowledge by evaluating two common surgical techniques to determine which may lead to better outcomes for patients undergoing TKA, a common orthopedic procedure, and reduce dissatisfaction as well as pain following operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 18
* Patients undergoing primary TKA for osteoarthritis

Exclusion Criteria:

* Patients undergoing revision TKA
* Any patients not undergoing TKA for non-OA diagnosis
* Adults unable to consent
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Pain Scale (VAS) | Before and after surgery at the 3 month, 6 month, and 12 month follow-ups
  The visual analog scale (VAS) is a tool used to measure pain. Patients will be asked to indicate their perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge .
Change in Oxford Knee Score (OKS) | Before and after surgery at the 3 month, 6 month, and 12 month follow-ups
  The Oxford Knee Score (OKS) is a 12-item patient-reported outcomes (PRO) specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty)
Change in Incidence of Pes bursitis | 3 weeks, 3 months, 6 months, and 12 months post-operatively.
  All patients will be seen post-operatively to monitor their progress and minimize risks, and the diagnosis of pes bursitis will be determined through clinical exam.

SECONDARY OUTCOMES:
Changes in Varus valgus knee assessment | 3 weeks, 3 months, 6 months, and 12 months post-operatively.
  This assessment checks the lateral and medial collateral ligaments (ligaments on either side of the knee joint that help in back and forth movement of knee). In this test, the study doctor will hold the patient's knee joint with one hand and the ankle joint with the other, and moves the patient's leg sideways to asses the ligaments.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Orthopaedics and Spine Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
At this time it will be an internal study with no sharing of de-identified patient information to third parties.